CLINICAL TRIAL: NCT06505044
Title: Effect of Moderate Intensity Aerobic Exercise Versus Resistance Exercise on Bone Density in Postmenopausal Diabetic Women
Brief Title: Effect of Aerobic Exercise Versus Resistance Exercise on Bone Density in Postmenopausal Diabetic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physical Therapy
Record Dates: First submitted 2024-07-02; First posted 2024-07-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind masking the patient was not be informed about the training group or the other group; they will be evaluated and trained at different places and times.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): 25 patients receive aerobic exercise attended the program of walking on a treadmill machine for eight weeks according to specific parameters, in addition to their usual daily calcium intake.
  Interventions: Procedure: aerobic exercise; Procedure: resistance exercise
- Group (B) (Active Comparator): 25 patients receive resisted exercise in addition to their usual daily calcium intake for 12 weeks.
  Interventions: Procedure: aerobic exercise; Procedure: resistance exercise

INTERVENTIONS:
Procedure: aerobic exercise — aerobic exercise.
  * Intensity: according to heart rate (60-75% of maximum heart rate) MHR=220-age.
  * Heart rate: determined by the sensor of a treadmill.
  * Duration: 40-50 min per session. Each session consisted of 5-10 minutes of warming up exercise on a treadmill without increasing speed or intensity and the same for the cooling down phase. There was 30 minutes of conditioning exercise including increasing the treadmill speed till reaching (60-75%) of the maximum heart rate.
  * Frequency: 3 times/week for 12 weeks in addition to their usual daily calcium intake.
Procedure: resistance exercise — resisted exercise program for 12 weeks

SUMMARY:
Osteoporosis is a significant public health issue, especially among postmenopausal women with diabetes, and its prevalence is increasing. This trial aims to determine the influence of moderate intensity aerobic exercise vs resistance exercise on bone mineral density among postmenopausal diabetic women.

DETAILED DESCRIPTION:
has diabetes. Postmenopausal Osteoporosis (PMO) is an increasingly serious metabolic bone disease in the world, which generally develops in middle-aged and elderly women and postmenopausal women, and it is characterized by low bone mass and microstructure degradation of bone tissues. there are complex pathophysiological effects between them: T2D directly affects bone metabolism and strength. Some antidiabetic drugs affect bone metabolism, and diabetes complications are related to the risk of falls and subsequent fractures. Patients with T2D have higher trabecular and lower cortical bone density, leading to lower bone intensity. Exercise is considered a highly relevant component in the prevention and treatment of osteoporosis and fracture reduction. Exercise greatly affects bone geometry as it increases periosteal apposition through increasing osteoblast formation. In addition to influencing bone mineral density, exercise can improve muscle function to potentially decrease fall risk through improved balance and strength.

The purpose of this study was to investigate the effect of moderate-intensity aerobic exercise versus resistance exercise on bone mineral density in postmenopausal diabetic women.

ELIGIBILITY:
Inclusion Criteria:

* Fifty women postmenopausal obese women
* (BMI) 30 -35 kg/m2
* their age ranges from 50 to 60 years old and
* complain of diabetic type 2 for 10 years ago.

Exclusion Criteria:

* women with renal or liver disease,
* cardiac or chest disease psychological problems,
* cognitive problems are excluded from the study.
* Any women who have therapeutic problems that will interfere with performing exercise or affection BMD will be excluded from this study.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The bone mineral density (BMD) | 3 months
  • Dual Energy X-ray Absorptiometry (DEXA). It was used to measure the bone mineral density (BMD) of the lumbar spine for each woman in both groups before and after the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Soad A. Mohamad, Minya, Egypt